CLINICAL TRIAL: NCT06161987
Title: Efficacy and Safety of Early Comprehensive Rehabilitation in Patients With ADHF, A Multicenter, Randomized, Controlled Trial.
Brief Title: EACH-ADHF: Early Comprehensive Rehabilitation in Patients With ADHF
Acronym: EACH-ADHF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lan Guo, Chief Physician of Cardiology, Director of the Department of Cardiac Rehabilitation, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-Q-2022-487-03
Record Dates: First submitted 2023-07-19; First posted 2023-12-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute decompensated heart failure; Early comprehensive rehabilitation; Inspiratory muscle training; Exercise training; KCCQ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation Intervention Group (Active Comparator): Comprehensive rehabilitation plan containing 18 sessions of a structured exercise and inspiratory muscle training program over 6 weeks (3 times per week).
  Interventions: Behavioral: Early comprehensive rehabilitation
- Attention Control (No Intervention): Conventional care with bi-weekly contact from study personnel.

INTERVENTIONS:
Behavioral: Early comprehensive rehabilitation — Patients randomized to the rehabilitation intervention group will be offered comprehensive rehabilitation plan containing 18 sessions of a structured outpatient-based exercise program over 6 weeks (3 times per week).
  Arms: Rehabilitation Intervention Group

SUMMARY:
EACH-ADHF: Early Comprehensive Rehabilitation in patients with ADHF study is a multi-center, parallel-group, randomized controlled trial designed to evaluate the effects of the early comprehensive rehabilitation including exercise and inspiratory muscle training, over a period of 6 weeks, on the quality of life of patients with ADHF.

DETAILED DESCRIPTION:
Guangdong Provincial People's Hospital will be the lead center, with an additional 8 hospitals designated as satellite centers for the study. To sum up, these centers will recruit a total of 140 consenting patients. Following informed consent and baseline testing, the participants will be randomized in a 1:1 fashion to receive a 6-week progressive, comprehensive exercise training and inspiratory muscle training or attention control.

The intervention group will receive an 6-week exercise program consisting of endurance, resistance, balance, mobility, and inspiratory muscle training. The comprehensive rehabilitation will begin during the patient's stay and continue to the outpatient clinic. The control group will receive usual care with bi-weekly contact from study personnel. The primary outcomes of the study are improvements in the summary score of KCCQ and PImax%pred, while secondary endpoints include the impact on physical function, cardiac function, psychological status, and major adverse cardiovascular events (MACE). Additionally, the study will also explore the effects of comprehensive rehabilitation on hospital readmission and mortality rates, with follow-up assessments planned up to 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80
2. At least one symptom of heart failure upon admission:

   Dyspnea at rest or with exertion, orthopnea, paroxysmal nocturnal dyspnea or exertional fatigue.
3. At least two of the signs of heart failure (HF):

   Distended jugular veins, enlarged cardiac silhouette, apex beat displacement, third heart sound, or increased jugular venous pressure/central venous pressure/pulmonary capillary wedge pressure.

   Pulmonary edema or pulmonary congestion (rales or chest X-ray/CT evidence of pulmonary congestion).

   Peripheral edema. Elevated B-type natriuretic peptide (>100 pg/ml) or elevated NT-proBNP (>300 pg/ml).
4. Able to independently perform basic activities of daily living before admission.
5. Able to complete the baseline assessment and initiate the specified treatment.
6. Able to walk 4 meters at the time of enrollment (assistive devices may be used).
7. Agree to participate in this study, sign a written informed consent form, and is willing to cooperate with follow-up.

Exclusion Criteria:

1. Acute heart failure caused by acute myocardial infarction.
2. Severe aortic valve stenosis.
3. Hemodynamic instability caused by poorly controlled arrhythmias.
4. Severe heart failure and high-degree atrioventricular block, and inadequate heart rate response to pacing during exercise.
5. Isolated pulmonary hypertension.
6. Poorly controlled symptomatic orthostatic hypotension.
7. Hypertrophic obstructive cardiomyopathy.
8. Stage 5 chronic kidney failure, defined as glomerular filtration rate <15 ml/(min·1.73m²) or requiring dialysis.
9. Undergoing screening tests with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than or equal to 5 times the upper limit of the normal range defined by the center.
10. Awaiting a heart transplant or ventricular assist device implantation within six months, or having received a heart transplant.
11. A history of chronic lung disease except for COPD, previous lung surgery, or diseases affecting lung function, such as scoliosis.
12. Late-stage diseases other than heart failure.
13. Any medical history that could potentially affect protocol compliance, such as severe mental disorders, severe cognitive impairment, substance abuse, or addiction.
14. Severe language, psychological, or physical disabilities that prevent their participation in the program.
15. Pregnant or lactating women, or those of childbearing potential who are unwilling or unable to use effective contraceptive measures.
16. Involved in other interventional clinical trials.
17. Patients deemed unfit for participation in this study by the researchers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Score of Quality of Life Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline and Week 6
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self-administered, 23-item questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life. All scores are represented on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Maximal Inspiratory Pressure as a Percentage of Predicted Value (PImax%pred) | Baseline and Week 6
  Participants will tries their best to exhale to the residual position, and then inhale as much as possible for 2~3 seconds to measure PImax and the percentage of PImax%pred

SECONDARY OUTCOMES:
Score of Short Physical Performance Battery (SPPB) | Baseline and Week 6
  The SPPB measures physical function using 3 components: standing balance with progressively narrow base of support, usual gait speed over 4 meters, and time to complete 5 chair rises. The total score ranges from 0 to 12, with higher scores indicating better physical function.
Score of Frailty | Baseline and Week 6
  Patients were classified as frail if they met three or more of the following criteria: weak grip strength, physical exhaustion, slowness, low physical activity and unintentional weight loss.
Pulmonary Function | Baseline and Week 6
  Measurements of forced vital capacity and forced expiratory volume in 1 s were obtained with a computerized spirometer.
Rate of All-Cause Rehospitalization | Month 6
  Number of all-cause rehospitalizations 6 months from hospital discharge.

OTHER OUTCOMES:
Score of Quality of Life Measured by Short Form 12 Item Questionnaire (SF-12) | Baseline and Week 6
  The SF-12 is a quality of life assessment with 2 component scores (Physical Composite Score and Mental Composite Score) ranging 0-100 with higher scores indicating better health status.
Score of Anxiety | Baseline and Week 6
  Anxiety is assessed by General Anxiety Disorder-7. Score ranges from 0 to 21 points, with higher scores indicating more severe anxiety.
Score of Depression | Baseline and Week 6
  Depression is assessed by Patient Health Questionnaire-9. Score of Patient Health Questionnaire-9 ranges from 0 to 27 points, with higher scores indicating more severe mood depression.
Left ventricular ejection fraction (LVEF) | Baseline and Week 6
  Using Echocardiography to assess the left ventricular ejection fraction (LVEF)
Left ventricular end-diastolic volume (LVEDV) | Baseline and Week 6
  Using Echocardiography to assess the left ventricular end-diastolic volume (LVEDV)
Left ventricular end-systolic volume (LVESV) | Baseline and Week 6
  Using Echocardiography to assess the left ventricular end-systolic volume (LVESV)
Rate of All-cause Rehospitalizations | Month 3, 6
  Number of all-cause rehospitalizations at 3 and 6 months from hospital discharge.
Rate of All-cause Composite Rehospitalization and Death | Month 3, 6
  Composite number of all-cause rehospitalizations and death at 3 and 6 months from hospital discharge.
The concentration of N-Terminal Pro-Brain Natriuretic Peptide （BNP/NT-proBNP） | Baseline and Week 6
  The concentration of N-Terminal Pro-Brain Natriuretic Peptide （BNP/NT-proBNP）
Incidence of adverse events and serious adverse events | Month 3, 6
  Incidence of adverse events and serious adverse events at 3 and 6 months from hospital discharge.
Incidence of Cardiovascular-related Composite Rehospitalization and Death | Month 3, 6
  Composite number of cardiovascular-related rehospitalizations and death at 3 and 6 months from hospital discharge.
Proteomics analysis | Baseline and Week 6
  Two 5ml tubes of blood were drawn at baseline and at 6 weeks, and a centrifuge was used to separate serum, plasma, and blood cells for mechanistic exploration.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitzman DW, Whellan DJ, Duncan P, Pastva AM, Mentz RJ, Reeves GR, Nelson MB, Chen H, Upadhya B, Reed SD, Espeland MA, Hewston L, O'Connor CM. Physical Rehabilitation for Older Patients Hospitalized for Heart Failure. N Engl J Med. 2021 Jul 15;385(3):203-216. doi: 10.1056/NEJMoa2026141. Epub 2021 May 16. PMID 33999544
- [Background] Mudge AM, Denaro CP, Scott AC, Meyers D, Adsett JA, Mullins RW, Suna JM, Atherton JJ, Marwick TH, Scuffham P, O'Rourke P. Addition of Supervised Exercise Training to a Post-Hospital Disease Management Program for Patients Recently Hospitalized With Acute Heart Failure: The EJECTION-HF Randomized Phase 4 Trial. JACC Heart Fail. 2018 Feb;6(2):143-152. doi: 10.1016/j.jchf.2017.11.016. PMID 29413370
- [Background] Reeves GR, Whellan DJ, Duncan P, O'Connor CM, Pastva AM, Eggebeen JD, Hewston LA, Morgan TM, Reed SD, Rejeski WJ, Mentz RJ, Rosenberg PB, Kitzman DW; REHAB-HF Trial Investigators. Rehabilitation Therapy in Older Acute Heart Failure Patients (REHAB-HF) trial: Design and rationale. Am Heart J. 2017 Mar;185:130-139. doi: 10.1016/j.ahj.2016.12.012. Epub 2016 Dec 28. PMID 28267466
- [Background] Laoutaris ID, Piotrowicz E, Kallistratos MS, Dritsas A, Dimaki N, Miliopoulos D, Andriopoulou M, Manolis AJ, Volterrani M, Piepoli MF, Coats AJS, Adamopoulos S; ARISTOS-HF trial (Aerobic, Resistance, InSpiratory Training OutcomeS in Heart Failure) Investigators. Combined aerobic/resistance/inspiratory muscle training as the 'optimum' exercise programme for patients with chronic heart failure: ARISTOS-HF randomized clinical trial. Eur J Prev Cardiol. 2021 Dec 29;28(15):1626-1635. doi: 10.1093/eurjpc/zwaa091. PMID 33624071
- [Background] Wu L, Li J, Chen L, Xue M, Zheng Y, Meng F, Jiang H, Shi Z, Zhang P, Dai C. The Efficacy and Safety of Phase I Cardiac Rehabilitation in Patients Hospitalized in Cardiac Intensive Care Unit With Acute Decompensated Heart Failure: A Study Protocol for a Randomized, Controlled, Clinical Trial. Front Cardiovasc Med. 2022 Mar 8;9:788503. doi: 10.3389/fcvm.2022.788503. eCollection 2022. PMID 35350537
- [Background] McNallan SM, Chamberlain AM, Gerber Y, Singh M, Kane RL, Weston SA, Dunlay SM, Jiang R, Roger VL. Measuring frailty in heart failure: a community perspective. Am Heart J. 2013 Oct;166(4):768-74. doi: 10.1016/j.ahj.2013.07.008. Epub 2013 Sep 17. PMID 24093859
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Spertus JA, Jones PG, Kim J, Globe D. Validity, reliability, and responsiveness of the Kansas City Cardiomyopathy Questionnaire in anemic heart failure patients. Qual Life Res. 2008 Mar;17(2):291-8. doi: 10.1007/s11136-007-9302-5. Epub 2007 Dec 29. PMID 18165909
- [Background] Takada S, Kondo T, Yasunaga M, Watanabe S, Kinoshita H, Fukuhara S, Yamamoto Y. Early rehabilitation in older patients hospitalized with acute decompensated heart failure: A retrospective cohort study. Am Heart J. 2020 Dec;230:44-53. doi: 10.1016/j.ahj.2020.09.009. Epub 2020 Sep 19. PMID 32956621